CLINICAL TRIAL: NCT02292394
Title: A Study of Randomized Controlled Dismantling of a Brief Telephone Psychological Intervention Applied to Informal Caregivers With Depressive Symptoms
Brief Title: Brief Telephone Psychological Intervention for Depressive Symptoms in Caregivers
Acronym: RCDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Ministry of Work and Welfare - Xunta de Galicia (Other Government)
Responsible Party: Principal Investigator, Fernando Lino Vázquez González, Associate Professor [Tenured Professor], University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSI2012-37396
Record Dates: First submitted 2014-11-06; First posted 2014-11-17 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Depression
Keywords: Depression; Depressive symptoms; Prevention; Caregivers; Telephone intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multicomponent Cognitive Behavioral Telephone Intervention (Experimental): In this study, we will apply a telephone intervention that is a modified version of a brief prevention intervention for depressed caregivers that previously was applied in person in a group format during five 90-minute sessions (Vazquez et al., 2014). During the intervention, participants will be trained in various behavioral and cognitive abilities such as increasing pleasant activities, self-reinforcement, relaxation techniques, assertive communication, strategies to increase social contacts and social skills, and strategies to increase positive thoughts and decrease depressive ones.
  Interventions: Behavioral: Multicomponent Cognitive Behavioral Telephone Intervention
- Telephone Intervention Pleasant Activities (Experimental): This intervention is also a modified version of a protocol described by Vazquez et al. (2014). However, in this case, we will specifically focus on the behavioral activation components of the multicomponent cognitive-behavioral telephone intervention. This intervention will also be structured in groups and administered by phone in five 90-minute sessions.
  Interventions: Behavioral: Telephone Intervention Pleasant Activities
- Usual care (No Intervention): Individuals assigned to this group will receive no intervention or material, but they will have unrestricted access to any routine medical or psychological care that they might want to seek to treat depressive symptoms. The use of such treatments will be recorded.

INTERVENTIONS:
Behavioral: Multicomponent Cognitive Behavioral Telephone Intervention
  Arms: Multicomponent Cognitive Behavioral Telephone Intervention
Behavioral: Telephone Intervention Pleasant Activities
  Arms: Telephone Intervention Pleasant Activities

SUMMARY:
Caring for dependent persons can give rise to depression in non-professional caregivers, placing a burden on health care services and threatening the quality of the care dispensed to the dependent. Unfortunately, the ability of these patients to attend therapy sessions is often limited precisely by their role as caregivers. Preventive measures that are accessible to caregivers are thus called for. The primary aim of this project is to evaluate the efficacy of telephonic administration of a brief indicated preventive psychological intervention for depression that in previous work proved effective when administered in person in group sessions. With a view to optimizing resource usage by maximizing interventional efficacy, the secondary aim is to determine the contribution to overall efficacy of that part of the intervention that consists in increasing pleasant activities. To these ends, some 180 informed, consenting caregivers satisfying appropriate criteria for inclusion in the study will be randomized to one of three interventions (≈ 60 participants per intervention): the full cognitive-behavioural programme; a program focused only on the component of pleasant activities; or a usual care condition. Both programmes will be administered in five 90 minute sessions by audio tele-conference. All sessions will be recorded for verification of adherence to the intervention protocols. Participants will be re-evaluated at the end of their intervention (when participant satisfaction with the cognitive-behavioural programmes will also be assessed) and also 1, 3, 6 and 12 months later; all evaluations will be performed by trained interviewers who will be blind to the aims of the study, the interventions employed, and the group to which any given participant belongs. Analyses of these evaluations will compare the short- and long-term efficacies of the three groups. Factors that mediate participant improvement or predict results will also be investigated, and the cost-effectiveness of the interventions will be estimated.The central hypothesis of the proposed study is that a multicomponent cognitive-behavioral telephone intervention and a protocol assessing participation in pleasant activities will both significantly reduce the incidence of depression and depressive symptoms compared to a control group with usual care immediately after treatment and at 1-, 3-, 6-, and 12-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Serves as an informal caregiver for dependent family member
* Dependence is recognized by the Xunta de Galicia
* Commitment to participate in all assessments
* A CES-D score ≥16
* Not suffering from a depressive episode
* Provides informed consent
* Has a telephone

Exclusion Criteria:

* Having received psychological or pharmacological treatment in the previous 2 months
* To present other conditions that may act as confounders (e.g., symptoms due to substance use)
* Presenting serious psychological or medical disorders that require immediate intervention (e.g., suicidal ideation) or prevent study implementation (e.g., significant cognitive impairment, severe hearing impairment)
* The dependent has a serious or terminal prognosis for the next 14 months
* Planning a change of address or institutionalization of the family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline Major depressive episode to post-treatment (6 weeks), and follow-ups at 1, 3, 6 and 12 months | Pre- and post-intervention (6 weeks) with follow-ups at 1, 3, 6, and 12 months
  The presence of a major depressive episode will be assessed with the Structured Clinical Interview for Axis I Disorders from the Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV Clinical Version (Structured Clinical Interview for DSM-IV, Clinician Version [SCID-CV]; First, Spitzer, Gibbon and Williams, 1997/1999). This is a semi-structured interview that provides a DSM-IV diagnosis and must be administered by a clinician. It consists of six modules of diagnostic interviews: mood episodes, psychotic symptoms, psychotic disorders, mood disorders, substance use disorders, anxiety disorders, and other disorders. The SCID-CV has good test-retest reliability and adequate reliability for psychiatric patients (kappa index = 0.61)

SECONDARY OUTCOMES:
Change from baseline depressive symptomatology to post-treatment (6 weeks), and follow-ups at 1, 3, 6 and 12 months | Pre- and post-intervention (6 weeks) with follow-ups at 1, 3, 6, and 12 months
  Depressive symptoms as measured by the Center for Epidemiological Studies Depression Scale [CES-D] (Radloff, 1977; Spanish version of Vazquez, White, and Lopez, 2007). This 20-item scale is self-administered and assesses depressive symptoms. The person evaluates each item based on how often they have experienced it in the last week using a Likert scale with four response options ranging from 0 (rarely or none of the time) to 3 (most of the time). The total score ranges from 0 to 60, and higher scores correspond to greater depressive symptomatology. Internal consistency (Cronbach's alpha) of the scale ranges from .85 and .90, with .89 for the Spanish version (Vazquez et al., 2007 and 2014).

OTHER OUTCOMES:
Socio-demographic characteristics | Pre-intervention
  Socio-demographic characteristics were collected via the Care Characteristics and Status of Caregiver questionnaire that was developed in a previous study (Vazquez et al., 2014). The data of caregivers (sex, age, marital status, number of children, social class, family monthly income per household, level of education, main occupation, province and area of residence), the care situation, health of the caregiver, and contact information (landline home phone)
Change from baseline Automatic negative thoughts to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  The occurrence of automatic negative thoughts will be assessed through the 30-item Automatic Negative Thoughts Questionnaire (ATQ-N, Hollon and Kendall, 1980). The subject must indicate the frequency for which a number of thoughts have suddenly arisen in their mind over the last week on a five-point scale from 1 (never) to 5 (always). Scores range between 30 and 150, and there is a direct relationship between the score and the frequencies of certain types of thoughts, with a higher score indicating more negative thoughts experienced by the subject. The internal consistency for the ATQ-N subscale is .96.
Change from baseline Behavioral activation to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  To assess behavioral activation, we will use the Environmental Reward Observation Scale (EROS, Armento and Hopko, 2007; Spanish version Barraca and Pérez-Álvarez, 2010). It is a self-administered 10-item scale that assesses the degree of positive reinforcement contingent on the response received from the media. Each item is evaluated based on the degree to which the individual believes applies to them, according to a Likert scale with four response options ranging from 1 (strongly disagree) to 4 (strongly agree), with higher scores indicating a greater degree of positive reinforcement. The total score ranges from 10 to 40. The Spanish version of EROS is reliable (Cronbach's alpha = .86) and valid (high correlations with the BDI-II, BADS, STAI-S/R, AAQ, significant differences between participants and non-clinical subjects).
Change from baseline Social contacts to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  To evaluate the participants' weekly social contacts we will use the Register of Social Networking (developed and used in the previous study by Vazquez et al., 2014) that asks the participants to report the number of people they had daily contact with.
Change from baseline Self-efficacy to post-treatment (6 weeks) | Pre- and post-intervention (6 weeks)
  Self-efficacy will be evaluated with the 10-item version of the General Self-Efficacy Scale (GSES, Jerusalem and Schwarzer, 1992; Spanish version Baessler and Schwarzer, 1996). This self-administered 10-item scale was designed to assess the feeling of personal competence to deal with difficult life situations. Each item is evaluated based on the degree to which the subject believes that the statement about their ability to solve problems is true on a Likert 4-point scale ranging from 1 (false) to 4 (true). Higher scores indicate a greater expectation of self-efficacy. Internal consistency for the Spanish version, estimated by Cronbach's alpha was .81.
Dropout and treatment adherence | During the intervention sessions (5 weeks)
  We will construct a registry of dropouts from each group to assess their response to the interventions over the duration of the study. In addition, treatment adherence will be assessed by recording the number of meetings each caregiver attends and whether they complete homework assignments.
Satisfaction with the service received | Post-intervention (6 weeks)
  Participant satisfaction with the service received will be evaluated upon intervention completion. We will use the Client Satisfaction Questionnaire ([CSQ-8]; Larsen, Attkisson, Hargreaves, and Nguyen, 1979; Spanish version Vazquez, Torres, and Otero, 2009). It is an 8-item scale with 4 possible answers and a final ranking score ranging from 8 to 32, where a higher score implies greater satisfaction with the service received. It is a widely used tool with an internal consistency between .83 and .93 (Attkisson and Greenfield, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L. Vázquez González, Associate Professor, Principal Investigator — University of Santiago de Compostela
Locations (1):
- Depressive Disorders Unit. School of Psychology. University of Santiago de Compostela., Santiago de Compostela, Galicia/A Coruña, Spain

REFERENCES:
- [Background] Armento ME, Hopko DR. The Environmental Reward Observation Scale (EROS): development, validity, and reliability. Behav Ther. 2007 Jun;38(2):107-19. doi: 10.1016/j.beth.2006.05.003. Epub 2006 Dec 12. PMID 17499078
- [Background] Attkisson CC; Greenfield TK. The UCSF Client Satisfaction Scales: I. The Client Satisfaction Questionnaire-8. In Maruish ME, editor, The use of psychological testing for treatment planning and outcomes assessment. 3rd ed. Volume 3. Mahwah, NJ: Lawrence Erlbaum Associates; 2004. p. 799-811.
- [Background] Baessler J; Schwarzer R. Evaluación de la autoeficacia: Adaptación española de la escala de Autoeficacia General. Anxiety & Stress 1996; 2: 1-8.
- [Background] Barraca J; Pérez-Álvaro M. Adaptación española del Environmental Reward Observation Scale (EROS). Anxiety & Stress 2010; 16: 95-107.
- [Background] First MB; Spitzer RL; Gibbon M; Williams, JBW Structured Clinical Interview for DSM-IV axis I disorders (SCID). New York: New York State Psychiatric Institute, Biometrics Research; 1997.
- [Background] Hollon SD; Kendall PC. Cognitive self-statements in depression: development of an Automatic Thought Questionnaire. Cognitive Ther Res 1980; 4: 383-395.
- [Background] Jerusalem M; Schwarzer R. Self-efficacy as a resource factor in stress appraisal processes. In Schwarzer R, editor. Self-efficacy: Thought control of action. Washington, DC: Hemisphere; 1992. p. 195-213.
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Radloff LS. A CES-D scale: a self-report depression scale for research in the general population. Appl Psychl Meas 1977; 1: 385-401.
- [Background] Vazquez FL, Blanco V, Lopez M. An adaptation of the Center for Epidemiologic Studies Depression Scale for use in non-psychiatric Spanish populations. Psychiatry Res. 2007 Jan 15;149(1-3):247-52. doi: 10.1016/j.psychres.2006.03.004. Epub 2006 Dec 1. PMID 17141880
- [Background] Vázquez FL; Hermida E; Torres A; Otero P; Blanco V; Díaz O. Eficacia de una intervención preventiva cognitivo conductual en cuidadoras con síntomas depresivos elevados. Behav Psychol 2014; 22: 77-94.
- [Background] Vázquez FL; Torres A; Otero P. CSQ-8 Castilian (TMS.047). Disponible en http://www.CSQscales.com; 2009.
- [Derived] Vazquez FL, Torres A, Diaz O, Otero P, Blanco V, Hermida E. Protocol for a randomized controlled dismantling study of a brief telephonic psychological intervention applied to non-professional caregivers with symptoms of depression. BMC Psychiatry. 2015 Nov 23;15:300. doi: 10.1186/s12888-015-0682-8. PMID 26597295